CLINICAL TRIAL: NCT07013747
Title: A Phase 1/2, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety, Efficacy and Immunogenicity of an Acne mRNA Vaccine Candidate in Participants With Mild Acne
Brief Title: Study to Evaluate Safety, Efficacy and Immunogenicity of Acne mRNA Vaccine in Participants With Mild Acne
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VBE00009; 2025-520677-39 (Registry Identifier: CTIS); U1111-1315-4645 (Registry Identifier: ICTRP)
Record Dates: First submitted 2025-06-02; First posted 2025-06-10 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Acne
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Intervention Model Description: This study will consist of a Core Study followed by an optional Long-Term Extension. Core Study will include a Sentinel Cohort and a Main Cohort, with the Sentinel Cohort assessing the safety in a stepwise manner.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Core Study:
  Sentinel Cohort: modified double-blind
  * Investigators, participants, laboratory personnel will be blinded
  * Clinical site staff preparing/administering the study vaccines will be unblinded
  * Sponsor study staff involved in early safety data reviews (ESDRs) will be unblinded at the time of the ESDR Main Cohort: modified double-blind
  * Investigators, participants, laboratory personnel and Sponsor study staff will be blinded
  * Clinical site staff preparing/administering the study vaccines will be unblinded
  * Sponsor staff involved in the Internal Firewall Committee will be unblinded at the time of the interim analysis
  Long-term Extension:
  Sentinel and Main Cohorts: double-blind
  • Investigators, participants, laboratory personnel and Sponsor study staff will be blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Sentinel Cohort Arm 1 (Experimental): Participants will receive 2 Acne mRNA Vaccine injections
  Interventions: Biological: Acne mRNA vaccine
- Sentinel Cohort Arm 2 (Placebo Comparator): Participants will receive 2 Placebo injections
  Interventions: Other: Placebo
- Main Cohort Arm 1 (Experimental): Participants will receive 2 Acne mRNA Vaccine injections
  Interventions: Biological: Acne mRNA vaccine
- Main Cohort Arm 2 (Placebo Comparator): Participants will receive 2 Placebo injections
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Acne mRNA vaccine — Pharmaceutical form: suspension for injection Route of administration: intramuscular
  Arms: Main Cohort Arm 1; Sentinel Cohort Arm 1
Other: Placebo — Pharmaceutical form: liquid solution for injection Route of administration: intramuscular
  Arms: Main Cohort Arm 2; Sentinel Cohort Arm 2

SUMMARY:
The purpose of the VBE00009 study is to evaluate the safety, efficacy and immunogenicity of 2 administrations of the Acne mRNA vaccine candidate at single dose level in participants aged 18 to 45 years with mild acne. This study will consist of a Core Study followed by an optional Long-Term Extension (LTE). Core Study will include a Sentinel Cohort and a Main Cohort, with the Sentinel Cohort assessing the safety in a stepwise manner. If the participants consent to the LTE, they will be followed up for an additional 30 months after the last planned visit in the Core Study, to assess the long term effects of the vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, and laboratory tests as judged by the investigator
* Clinical diagnosis of mild facial acne vulgaris with:

  * IGA score of mild (grade 2 on the 5-grade IGA scale) AND
  * between 10 to 24 non-inflammatory lesions (ie, open and closed comedones) AND
  * between 5 to 19 inflammatory lesions (ie, papules and pustules) AND
  * no nodulocystic lesions (ie, nodules and cysts)

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within 6 months prior to the first study intervention administration; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
* Known systemic hypersensitivity to any of the study intervention components (eg, polyethylene glycol [PEG], polysorbate); history of a life-threatening reaction to the study interventions used in the study or to a product containing any of the same substances; any allergic reaction (eg, anaphylaxis) after administration of mRNA coronavirus disease 2019 (COVID 19) vaccine
* Previous history of myocarditis and/or pericarditis and/or myopericarditis
* Skin pathology or condition that, in the investigator's opinion, could interfere with the evaluation of the study intervention or requires use of interfering topical, systemic, or surgical therapy
* Excessive facial hair, facial tattoos, facial skin disorders, skin reactions that may interfere with the study assessments in the investigator's opinion (including - but not limited to - actinic keratosis, eczema, psoriasis, seborrheic dermatitis, rosacea, acute or recent sunburn) or skin infection
* Receipt of immune globulins, blood or blood-derived products in the past 3 months
* Self-reported or documented seropositivity for human immunodeficiency virus (HIV), hepatitis B virus, or hepatitis C virus

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-07-03 (Actual); Primary Completion 2029-06-19 (Estimated); Study Completion 2029-06-19 (Estimated)

PRIMARY OUTCOMES:
Core Study - Sentinel Cohort Arm 1 and 2: Number of participants with unsolicited systemic adverse events (AEs) | In 30 minutes after each administration
Core Study - Sentinel Cohort Arm 1 and 2: Number of participants with solicited injection site and systemic reactions | Up to 7 days after each administration
  pre-listed in the participant diary [PDi] and in the case report form [CRF]
Core Study - Sentinel Cohort Arm 1 and 2: Number of participants with unsolicited AEs reported | Up to 28 days after each administration
Core Study - Sentinel Cohort Arm 1 and 2: Number of participants with medically attended adverse events (MAAEs) | Up to 6 months after each administration
Core Study - Sentinel Cohort Arm 1 and 2: Number of participants with AEs of special interest (AESIs) | Up to 6 months after each administration
Core Study - Sentinel Cohort Arm 1 and 2: Number of participants with serious AEs (SAEs) | Up to 6 months after each administration
  Presence of all SAEs
Core Study - Sentinel Cohort Arm 1 and 2: Number of participants with out-of-range biological test results | Through 7 days after administration (Day 08)
  Presence of out-of-range biological test results (including shift from baseline values)
Core Study - Main Cohort Arm 1 and 2: Percentage change from baseline (Day 01) in the number of inflammatory acne lesions on face | At 2 months post last administration
Core Study - Main Cohort Arm 1 and 2: Percentage change from baseline (Day 01) in the number of non-inflammatory acne lesions on face | At 2 months post last administration
Long-Term Extension - Sentinel and Main Cohort Arm 1 and 2: Number of participants with serious adverse events (SAEs) and adverse events of special interest (AESIs) | Up to 38 months after first administration
  Presence of all SAEs and AESIs

SECONDARY OUTCOMES:
Core Study - Sentinel and Main Cohort Arm 1 and 2: Vaccine-antigen-specific serum antibody titers | From baseline (Day 01) to 6 months post last administration
Core Study - Main Cohort Arm 1 and 2: Absolute change from baseline (Day 01) in the number of inflammatory acne lesions on face | At 1 month post first administration to 6 months post last administration
Core Study - Main Cohort Arm 1 and 2: Percentage change from baseline (Day 01) in the number of inflammatory acne lesions on face | At 1 month post first administration to 6 months post last administration
Core Study - Main Cohort Arm 1 and 2: Absolute change from baseline (Day 01) in the number of non-inflammatory acne lesions on face | At 1 month post first administration to 6 months post last administration
Core Study - Main Cohort Arm 1 and 2: Percentage change from baseline (Day 01) in the number of non-inflammatory acne lesions on face | At 1 month post first administration to 6 months post last administration
Core Study - Main Cohort Arm 1 and 2: Number of participants with unsolicited systemic adverse events (AEs) | In 30 minutes after each administration
Core Study - Main Cohort Arm 1 and 2: Number of participants with solicited injection site and systemic reactions | Up to 7 days after each administration
  pre-listed in the participant diary [PDi] and in the case report form [CRF]
Core Study - Main Cohort Arm 1 and 2: Number of participants with unsolicited AEs reported | Up to 28 days after each administration
Core Study - Main Cohort Arm 1 and 2: Number of participants with medically attended adverse events (MAAEs) | Up to 6 months after each administration
Core Study - Main Cohort Arm 1 and 2: Number of participants with AEs of special interest (AESIs) | Up to 6 months after each administration
Core Study - Main Cohort Arm 1 and 2: Number of participants with serious AEs (SAEs) | Up to 6 months after each administration
  Presence of all SAEs
Core Study - Main Cohort Arm 1 and 2: Number of participants with out-of-range biological test results | Through 7 days after administration (Day 08)
  Presence of out-of-range biological test results (including shift from baseline values)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Encino Research Center- Site Number : 8400008, Encino, California
  - Moore Clinical Research - Brandon- Site Number : 8400007, Brandon, Florida
  - Encore Research Group-Jacksonville Center for Clinical Research- Site Number : 8400006, Jacksonville, Florida
  - DelRicht Research- Site Number : 8400003, New Orleans, Louisiana

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: VBE00009 Plain Language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=26705&tenant=MT_SNY_9011